CLINICAL TRIAL: NCT03427866
Title: A Phase II Study of Ruxolitinib Pre-, During- and Post-Hematopoietic Stem Cell Transplantation for Patients With Primary or Secondary Myelofibrosis.
Brief Title: Ruxolitinib Pre-, During- and Post-HSCT for Patients With Primary or Secondary Myelofibrosis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Gabriela Hobbs, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-569
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ruxolitinib Eligible pre-HSCT (Experimental): * Ruxolitinib will be taken orally at a fixed dose twice every day
  * Dosing will be continuous, with a new cycle scheduled to start every 28 days.
  * There will be no break in dosing between cycles
  * Ruxolitinib can be administered with or without food.
  Interventions: Drug: Ruxolitinib
- Ruxolitinib Not Eligible pre-HSCT (Experimental): * Ruxolitinib will be taken orally at a fixed dose twice every day after transplant
  * Dosing will be continuous, with a new cycle scheduled to start every 28 days.
  * There will be no break in dosing between cycles
  * Ruxolitinib can be administered with or without food.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib is a medication that blocks certain proteins called tyrosine kinases. Specifically, it blocks tyrosine kinases called JAK2. The JAK2 pathway is over active in the disease, acute myeloid leukemia.
  Other Names: Jakafi

SUMMARY:
This research study is studying a drug called Ruxolitinib as a possible treatment for Myelofibrosis.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has approved Ruxolitinib as a treatment option for this disease.

This study examines two different cohorts of participants:

* Cohort 1: Participants who are eligible for Ruxolitinib therapy before transplant, based on their platelet counts. These participants will receive their first dose of the study drug between 2 and 6 months before HCT.
* Cohort 2: Participants who are not eligible for Ruxolitinib therapy pre-treatment based on their platelet counts. These participants will receive their first dose of Ruxolitinib 1 week before the conditioning period.

Ruxolitinib is a medication that blocks certain proteins called tyrosine kinases. Specifically, it blocks tyrosine kinases called JAK2. Many cancers have over active "cell signaling." What this means is that certain functions in the cancer cells never turn off and this makes them grow in an uncontrolled way. Ruxolitinib, shuts down the pathway that depends on the JAK2 tyrosine kinases. The JAK2 pathway is over active in the participant's disease, acute myeloid leukemia. The exact way ruxolitinib does this is not yet clear but it may have to do with its ability to block the JAK2 pathway since this pathway can also lead to inflammation in the body.

Ruxolitinib has also been shown to lower the rates of Graft-Versus-Host-Disease (GVHD), a complication of transplant. GVHD is a disease that occurs when the immune cells in transplanted donor tissue from your HCT attack the participant's own tissues and organs. There are two types of GVHD: acute and chronic. Acute GVHD generally occurs within 1 week to 3 months after your HCT and may affect your skin, intestines, and liver. Chronic GVHD begins later on and may affect the organs prone to acute GVHD complications, as well as the lungs, mucous membranes, or other organs.

There is also evidence that ruxolitinib is associated with reduced instances of enlarged spleen size after HCT. Enlarged spleens play a role in the engraftment rate after HCT, which is the rate at which donated tissue and your own tissue begin reproducing and growing together.

In this research study, the investigators are:

* assessing the efficacy (how well the study drug works) and tolerability of Ruxolitinib before, during, and after HCT.
* examining the rates of GVHD after HCT when ruxolitinib is administered.
* determining whether engraftment rates improve when ruxolitinib is given

ELIGIBILITY:
Inclusion Criteria:

* Participants must have pathologically confirmed primary myelofibrosis according to WHO criteria1 or secondary myelofibrosis as defined by the IWG-MRT criteria.19

  * Intermediate-2/ high-risk disease as per Dynamic IPSS (DIPSS) criteria2 (Appendix 1) OR
  * Intermediate-1 risk disease with one of the following additional unfavorable features known to impact the survival adversely
  * Red cell transfusion dependency2
  * Unfavorable Karyotype2
  * Platelet count ≤100 x 109/L
* Age 18-75
* Participants must be designated to undergo reduced intensity allogeneic peripheral blood (PB) or bone marrow (BM) hematopoietic stem cell transplantation. Consent will be obtained prior to admission for HCT.
* Participants who will undergo HCT from the following donor types are eligible:
* 5/6 or 6/6 (HLA-A, B, DR) matched related donor
* 7/8 or 8/8 (HLA-A, B, DR, C) matched unrelated donor. Matching in the unrelated setting must be at the allele level
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Life expectancy of greater than 3 months
* Able to give informed consent
* Off all MF-directed therapy at the time of enrollment, with the exception of ruxolitinib
* Additional Criteria for Cohort 1 Only:
* Patients are candidates for enrollment in cohort 1 if they have an indication for ruxolitinib based on splenomegaly or symptoms and are either on ruxolitinib already or going to start therapy with ruxolitinib.
* Patients that are on ruxolitinib may enroll in study as long as they are willing to remain on ruxolitinib during the study and have not lost response to ruxolitinib defined as an increase in >5 cm in spleen size from nadir. There is no minimum or maximum time requirement for time on ruxolitinib.
* Participants must have splenomegaly (defined by ultrasound or CT scan of the abdomen) or symptoms (demonstrated by the presence of 1 symptom score >5 or 2 symptom scores >3) related to myelofibrosis as measured by the myeloproliferative neoplasm symptom assessment form MPN-SAF (see Appendix F) and platelets >25/μL and hemoglobin >7/dL
* Additional Criteria Cohort 2 Only:
* Participants are ineligible for ruxolitinib - do not have splenomegaly or symptoms of myelofibrosis as defined by the MPN-SAF.

Or

* Participants failed ruxolitinib as defined by loss of response to therapy and
* No allergy to ruxolitinib in the past

Exclusion Criteria:

* Hypersensitivity to any JAK inhibitor
* Prior allogeneic transplant for any hematopoietic disorder
* Had accelerated phase or leukemic transformation (≥10% blasts in PB or BM any time prior to HCT)
* Active uncontrolled infection
* History of another malignancy within 5-years of date of except h/o basal cell or squamous cell carcinoma of skin or Polycythemia Vera or Essential Thrombocythemia
* Patients without normal organ function defined as follows:

  * AST (SGOT), ALT (SGPT) and Alkaline Phosphatase ≥ 3 × institutional Upper Limit of Normal (ULN)
  * Direct bilirubin >2.0 mg/dL
  * Adequate renal function as defined by calculated creatinine clearance≤60 mL/min (Cockcroft-Gault formula)
* Have a chronic or active infection that requires systemic antibiotics, antifungal or antiviral treatment
* Have current or a history of congestive heart failure New York Heart Association (NYHA) class 3 or 4, or any history of documented diastolic or systolic dysfunction (LVEF < 40%, as measured by MUGA scan or echocardiogram)
* Pregnancy at the time of enrollment
* Unable to give informed consent
* Have an uncontrolled intercurrent illness including, but not limited to, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects who require therapy with a strong CYP3A4 inhibitor prior to enrollment to this study
* Not able to take oral medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
GVHD free and relapse free survival at 1 year | 1 year
  The number of participants surviving after one year that have not experienced graft-versus host disease (GVHD) or relapse (GRFS rate)

SECONDARY OUTCOMES:
Progression Free Survival | 1 and 2 years
  Kaplan-Meier estimates of progression free survival (PFS) will be calculated, with patients without an event being censored at 1 and 2 years
Overall Survival | 1 and 2 years
  Overall survival is measured as the time from the hematopoietic stem cell transplantation (HSCT) until death. Participants without an event will be censored at the date of last contact.
Cumulative incidence of aGVHD | 6 months
  Cumulative incidence of grades II-IV and II-IV acute GVHD at 6 months after HSCT
Cumulative incidence of cGVHD | 1 and 2 years
  Cumulative incidence of moderate to severe chronic GVHD at 1 year and 2 years after HSCT
Rate of Engraftment | 2 years
  Engraftment defined as ANC >500/ugx3 consecutive measurements and platelets of >20x10e9/L for three consecutive days.
Median time on ruxolitinib after HSCT as a measure of feasibility | 2 years
  The amount of time patients remain on ruxolitinib from transplant until discontinuation.
Toxicity rate | 2 years
  Cumulative incidence of treatment related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE 4). Early deaths from all other causes are considered a competing risk.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Hobbs, MD, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No